CLINICAL TRIAL: NCT01515826
Title: Evaluation of the Safety and Efficacy of VIGADEXA Ophthalmic Gel Compared to VIGADEXA Ophthalmic Solution in Preventing Inflammation and Infection Following Cataract Surgery
Brief Title: VIGADEXA Gel Compared to VIGADEXA Solution Following Cataract Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-10-013
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Cataracts
Keywords: Cataract surgery; Topical therapy; Prevention of inflammation; Inflammation of infection
MeSH Terms: conditions — Cataract | interventions — Moxifloxacin; dexamethasone 21-phosphate; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VIGADEXA Gel (Experimental): VIGADEXA ophthalmic gel topically administered TID to the operative eye starting the day before surgery, continuing on the day of surgery, and for 15 days following surgery.
  Interventions: Drug: Moxifloxacin 0.5%/Dexamethasone Phosphate 0.075% Ophthalmic Gel (VIGADEXA Gel)
- VIGADEXA Solution (Active Comparator): VIGADEXA ophthalmic solution topically administered QID to the operative eye starting the day before surgery, continuing on the day of surgery, and for 15 days following surgery.
  Interventions: Drug: Moxifloxacin 0.5%/Dexamethasone Phosphate 0.1% Ophthalmic Solution (VIGADEXA Solution)

INTERVENTIONS:
Drug: Moxifloxacin 0.5%/Dexamethasone Phosphate 0.075% Ophthalmic Gel (VIGADEXA Gel) — One ribbon (approximately 1-1.5 cm) administered topically in the conjunctival sac of the study eye three times daily (TID), starting the day before surgery (Day -1) and continuing on the day of surgery and for 15 days following surgery.
  Other Names: FID 119149, VIGADEXA Gel
  Arms: VIGADEXA Gel
Drug: Moxifloxacin 0.5%/Dexamethasone Phosphate 0.1% Ophthalmic Solution (VIGADEXA Solution) — One drop administered topically in the conjunctival sac of the study eye four times daily (QID), starting the day before surgery (Day -1) and continuing on the day of surgery and for 15 days following surgery.
  Other Names: VIGADEXA Solution
  Arms: VIGADEXA Solution

SUMMARY:
The purpose of this study is to compare VIGADEXA (moxifloxacin 0.5%/dexamethasone phosphate 0.075%) ophthalmic gel to VIGADEXA (moxifloxacin 0.5%/dexamethasone phosphate 0.1%) ophthalmic solution in the prevention of postoperative inflammation and infection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Diagnosis of cataract with intention to undergo routine, uncomplicated cataract surgery.
* Able to understand and sign an informed consent form.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Glaucoma or ocular hypertension.
* Use of topical or systemic non-steroidal anti-inflammatory drugs (NSAIDs) within 14 days prior to surgery or planned use during the study. Low-dose acetylsalicylic acid (up to 100 mg/day) is allowed.
* Use of anti-bacterial, anti-viral, or anti-fungal agents or ocular medications within 30 days prior to enrollment in the study or during study, as specified by protocol.
* Secondary implantation or replacement of the intra-ocular lens (IOL) in the study eye.
* Planned use of contact lenses in the study eye during the study period.
* Cataract surgery in the contralateral eye within 30 days prior to the Screening Visit, or planned for the 3 weeks after the cataract surgery in the study eye.
* History of clinically significant trauma to the study eye within the past 12 months.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a score of 0 (<5 cells) for cells in the anterior chamber | Day 15 post-operative
  As assessed by the investigator during slit-lamp examination.
Percentage of patients with no clinically evidenced bacterial infection | Day 15 post-operative
  As assessed by the investigator during slit-lamp examination.

SECONDARY OUTCOMES:
Cells in the anterior chamber (study eye) | Day 15 post-operative
  As assessed by the investigator during slit-lamp examination.
Ocular pain (study eye) | Day 15 post-operative
  As assessed by the investigator during patient interview.
Inflammatory reaction (study eye) | Day 15 post-operative
  As assessed by the investigator during slit-lamp examination.